CLINICAL TRIAL: NCT06443437
Title: Effect of Bee-buzzy Vibrating Cold Application and Marionette Doll on Pain and Fear During Phlebotomy Among Preschool Children: A Randomized Controlled Study
Brief Title: Effect of Bee-buzzy Vibrating Cold Application and Marionette Doll on Pain and Fear During Phlebotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Hassan Khalf allah, lecturer, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: bee-buzzy&marionette doll
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Fear of Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group 1 (Experimental): children who will receive bee-buzzy vibrating cold application
  Interventions: Other: bee-buzzy vibrating cold application marionette doll
- study group 2 (Active Comparator): children who will receive marionette doll
  Interventions: Other: bee-buzzy vibrating cold application marionette doll
- control group (Other): children who will receive routine care
  Interventions: Other: Rotuine care

INTERVENTIONS:
Other: bee-buzzy vibrating cold application marionette doll — * Bee-buzzy will be attached to the arm of the preschool child (who is included in the bee-buzzy group) by the researchers, where the phlebotomy will be performed on the child. It reduces pain through its cold wings and vibration. It helps to distract attention during phlebotomy and reduces the feeling of pain and fear. Bee-buzzy will be tied 5 cm above the area from which blood will be drawn, and after waiting for 15 seconds, the nurse will perform a phlebotomy.
  * A marionette doll group; while the nurse is going to perform the phlebotomy operation on the preschool child, one of the researchers will try to distract the child by paly with marionette doll. The researchers will receive training in play therapy
  Other Names: marionette doll
  Arms: study group 1; study group 2
Other: Rotuine care — children in control group will receive routine hospital are
  Arms: control group

SUMMARY:
Non-pharmacological methods are often used as a creative strategy to reduce pain and fear in children during a painful procedure such as phlebotomy. In this context, external vibratory cold application and a marionette doll are a commonly used as non-pharmacological distraction method to reduce pain and fear. In the literature, there are studies with cold application, vibrating devices and a marionette doll in bee appearance therefor this study is aimed to evaluate the effect of bee-buzzy vibrating cold application and marionette doll on pain and fear during phlebotomy among preschool children.

DETAILED DESCRIPTION:
Pain is one of the negative experiences faced in pediatric patients due to various medical interventions and often causes fear and anxiety. Pain perception is affected by the child's age, cognitive development, communication skills, previous pain experiences, and pain beliefs. Severe and long-term pain resulting from interventions can cause behavioral and physiological problems. In this period, if the pain is not alleviated or eliminated with appropriate interventions, it may cause neurological and behavioral disorders in the future. Nurses are responsible for minimizing the pain felt by children exposed to painful interventions and helping them cope with it .

ELIGIBILITY:
Inclusion Criteria:

1. children and parents who agreed to participate in the study
2. children had successful phlebotomy in the first attempt.

Exclusion Criteria:

1. Children who are having a chronic disease
2. Mental disability or mental retardation
3. Taking analgesics in the last 24 hours
4. Undergone a surgical procedure,
5. Not having a successful phlebotomy on the first attempt,
6. The child and his/her family not being willing to participate in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
child pain | during phlebotomy
  Facial expression rating scale (Wong-Baker Faces Pain Rating Scale). The Facial Expression Rating Scale includes 6 facial expressions and is a scale that provides a rating between 0 and 10 (Conlon, 2009; Huguet et al., 2010). Facial expressions range from"0" a smiling "brutal" face, 1-2 "It hurts a little", 3-4 "It hurts a little more", 5-6 "It hurts even more", 7-8 "It hurts a lot", and 9-10 "It hurts worst". This scale does not require words or numerical values and is a reliable and valid measurement tool in the assessment of acute pain. With this scale, the child's pain will be evaluated and recorded by both the nurse who will perform the phlebotomy and the parent.

SECONDARY OUTCOMES:
child fear | during phlebotomy
  The "Children's Fear Scale" by McMurtry et al. (2011). This scale includes 5 different facial expressions. This scale is scored between 0 and 4 and it is stated to be a reliable and valid measurement tool in the evaluation of fear (McMurtry et al., 2011). The permission to use the scale was obtained by Binay and Bal Yılmaz (2019), and Turkish validity and reliability studies were conducted (Binay & Bal Yılmaz, 2019; Binay & Bal Yilmaz, 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Safaa R Osman, post doctor, Study Chair — Assiut university faculty of nursing; . Nahed T Mohamed, post doctor, Study Chair — Assiut university faculty of nursing; Amira H Abdelfatah, post doctor, Study Director — Assiut university faculty of nursing
Locations (1):
- Assiut university children hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yildirim BG, Gerceker GO. The Effect of Virtual Reality and Buzzy on First Insertion Success, Procedure-Related Fear, Anxiety, and Pain in Children during Intravenous Insertion in the Pediatric Emergency Unit: A Randomized Controlled Trial. J Emerg Nurs. 2023 Jan;49(1):62-74. doi: 10.1016/j.jen.2022.09.018. Epub 2022 Nov 12. PMID 36376127
- [Background] Wang Y, Guo L, Xiong X. Effects of Virtual Reality-Based Distraction of Pain, Fear, and Anxiety During Needle-Related Procedures in Children and Adolescents. Front Psychol. 2022 Apr 19;13:842847. doi: 10.3389/fpsyg.2022.842847. eCollection 2022. PMID 35519646
- [Background] Ugucu G, Akdeniz Uysal D, Guzel Polat O, Artuvan Z, Polat Kulcu D, Aksu D, Gulgun Altintas M, Cetin H, Orekici Temel G. Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: A randomized experimental study. J Pediatr Nurs. 2022 Jul-Aug;65:e107-e114. doi: 10.1016/j.pedn.2022.03.016. Epub 2022 Apr 8. PMID 35410736
- [Background] Turgut MA, Turkmen AS. The effect of lighted toy on reducing pain and fear during blood collection in children between 3 and 6 years: A randomized control trial. J Pediatr Nurs. 2023 May-Jun;70:111-116. doi: 10.1016/j.pedn.2023.02.009. Epub 2023 Mar 9. PMID 36905910
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Kuo HC, Pan HH, Creedy DK, Tsao Y. Distraction-Based Interventions for Children Undergoing Venipuncture Procedures: A Randomized Controlled Study. Clin Nurs Res. 2018 May;27(4):467-482. doi: 10.1177/1054773816686262. Epub 2016 Dec 30. PMID 28038497